CLINICAL TRIAL: NCT01465581
Title: A Prospective Trial of Division of the Filum Terminale for Neurogenic Bladder Dysfunction With a Normal Conus
Brief Title: Treatment of Neurogenic Incontinence by Surgery to Cut the Filum Terminale
Acronym: NICNOC
Status: Terminated | Type: Observational
Why Stopped: Insufficient patient accrual.
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 228683
Record Dates: First submitted 2011-10-26; First posted 2011-11-07 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2011-11

CONDITIONS: Neurogenic Incontinence; Dysfunctional Voiding
Keywords: incontinence; dysfunctional voiding; neurogenic bladder disturbance; filum terminale; spinal cord tethering; conus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurogenic incontinence: The target population of this study is children with primary or secondary daytime urinary incontinence, who have failed to improve adequately despite compliance with at least 6 months of standard medical therapy. These children will have abnormal urodynamics, a normal bladder ultrasound and an MR imaging showing that the conus of the spinal cord is at a normal position and that there is no other significant dysraphic lesion present.
  Interventions: Procedure: Division of the filum terminal

INTERVENTIONS:
Procedure: Division of the filum terminal — Division of the filum is performed through a 6cm incision over the lumbosacral junction that can be oriented either longitudinally or transversely - to be hidden beneath underclothes or swim wear. A single level laminectomy provides sufficient exposure. The dural opening can be as short as 1cm. Under the microscope the filum is identified visually and separated from lower sacral rootlets with the aid of microelectrode stimulation. When a segment of the filum has been excised and sent for laboratory examination, the dura is closed and reinforced with fibrin glue. The wound is closed in layers, and the patient is kept at bed rest horizontal for 2 nights to discourage CSF fistulization of the wound.

SUMMARY:
The target population of this study is children with primary or secondary daytime urinary incontinence, who have failed to improve adequately despite compliance with at least 6 months of standard medical therapy.

The study hypothesis is that patients who under go cutting the filum terminale - the string-like lower end of the spinal cord - will have improved bladder function at 6-month follow up.

Bladder function and its effects on quality of life will be measured before surgery and at 6-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary daytime urinary incontinence, persistent over at least 6 months of medical treatment.
* Abnormal urodynamic testing
* Normal conus on magnetic resonance imaging of the spine
* Dysfunctional Voiding Symptom Scale score greater than 6 for girls or greater than 9 for boys

Exclusion Criteria:

* Bladder outlet obstruction
* Bladder atony
* Congenital anorectal malformation
* Additional diagnoses independently associated with neurogenic bladder dysfunction
* Encephalopathy precluding reasonable expectation of attainment of continence
* Inability to comply with medical management
* Unwillingness to comply with initial or follow up urodynamic testing

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population of this study is children with primary or secondary daytime urinary incontinence, who have failed to improve adequately despite compliance with at least 6 months of standard medical therapy. These children will have abnormal urodynamics, a normal bladder ultrasound and an MR imaging showing that the conus medullaris of the spinal cord is at a normal position and that there is no other significant dysraphic lesion present. The entry criteria are designed to separate this very specific subset of patients from the much larger, more general group of children presenting for evaluation and management of incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Pediatric Enuresis Module to Assess Quality of Life | 6-month follow up

SECONDARY OUTCOMES:
Change from baseline in a 24-hour voiding log | 6-month follow up
Change from baseline in the Dysfunctional Voiding Symptom Scale | 6-month follow up
Change from baseline urodynamic testing | 6-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Piatt, MD, Principal Investigator — Alfred I. duPont Hospital for Children
Locations (1):
- A I duPont Hospital for Children, Wilmington, Delaware, United States